CLINICAL TRIAL: NCT06870318
Title: Nutrient Enrichment of Human Milk With Human and Bovine Milk-based Fortifiers for Very Preterm Infants: an Individual Participant Data Meta-analysis
Brief Title: Enrichment of Human Milk With Human and Bovine Milk-based Fortifiers for Very Preterm Infants: a Meta-analysis
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Umeå University (Other); Region Östergötland (Other)
Responsible Party: Principal Investigator, Deborah O'Connor, Senior Associate Scientist, The Hospital for Sick Children
Other Study IDs: 4784
Record Dates: First submitted 2025-02-03; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Human Milk Fortification; Very Low Birth Weight Baby; Human Milk Nutrition; Human Milk Feeding; Necrotizing Enterocolitis (NEC); Late Onset Neonatal Sepsis; Growth; Feeding Intolerance in Preterm; Infant Mortality
Keywords: Bovine based vs human milk based fortifiers; RCTs meta-analysis; Human Milk Fortifiers (HMF)
MeSH Terms: conditions — Enterocolitis, Necrotizing; Neonatal Sepsis; Infant Death | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Human milk-based multi-nutrient fortifiers (HMBF) group: Infants born VLBW fed exclusively with Human Milk (parent milk or pasteurized donor milk) fortified with HMBF
  Interventions: Other: No intervention; Observational study
- Bovine milk-based fortifiers (BMBF) group: Infants born VLBW fed exclusively with Human Milk (parent milk or pasteurized donor milk) fortified with BMBF
  Interventions: Other: No intervention; Observational study

INTERVENTIONS:
Other: No intervention; Observational study — OptiMoM-NForte is meta-analysis study (observational secondary use of data), the investigators will analyze data from the OptiMoM and NForte trials. No interventions form part of this study.

SUMMARY:
Research has shown that provision of mother's milk is the optimal way to feed very low birthweight (VLBW) infants. Many infants will require a supplement to mother's milk, pasteurized donor human milk (PDHM) compared to preterm formula is the most appropriate supplement as it has been shown to reduce the risk of necrotizing enterocolitis (NEC).

Most available evidence suggests neither mother's milk nor PDHM will meet the elevated nutritional requirements of VLBW infants without multi-nutrient fortification. Globally, the current standard of care is to use bovine protein-based nutrient fortifiers to meet these elevated nutrient requirements. Given the known benefits of mother's milk, the reduction in the risk of NEC with use of PDHM as a supplement, and the availability of human milk-based multi-nutrient fortifiers (HMBF), there has been considerable interest in the efficacy of HMBF over the less costly bovine milk-based fortifiers (BMBF).

This study is an analysis of individual participant data merged from randomized control trials that examined the efficacy of HMBF compared to BMBF during hospitalization, on the risk of death and severe morbidity or major feeding interruption. Participants of the trials included in the analyses were fed exclusively with human milk or a supplement of pasteurized donor human milk (PDHM).

Only two RCTs met this criteria -OptiMoM and the N-forte trial. In both studies the intervention aligned to commence upon randomization into the HMBF or BMBF groups. The difference between the OptiMoM and N-forte feeding protocols was that the later allowed for individualized fortification based on milk analysis whereas OptiMoM used standard fortification, predominant in Canada and globally.

For OptiMoM, the feeding intervention continued until infants were 84 days of age, discharge, or when the infant consumed ≥2 complete oral feeds daily. For N-forte trial, the feeding intervention ended when babies reached 34 weeks (zero days). Both studies followed participants and continued data collection if transferred to a level II NICU for convalescence (OptiMoM) or home care service followed closely by NICU nurses (N-forte) until discharge.

ELIGIBILITY:
Inclusion Criteria:

• Infant is a participant of the OptiMoM or the N-Forte trial.

Ages: 1 Hour to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants of the OptiMoM and N-Forte trial are VLBW infants fed exclusively Human Milk.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with composite of NEC (NEC II-III), culture-proven late-onset sepsis and mortality. | From study day 1 through hospitalization, approximately 60 days.
  The first primary outcome is a binary (yes/no) composite of NEC (NEC II-III), culture-proven late-onset sepsis and mortality.
Percentage of infants with an interruption in enteral feeding. | Through feeding intervention, approximately 50 days.
  The second primary outcome is the percentage of infants with an interruption in enteral feeding after commencement of the intervention (e.g. Study Day 1), unrelated to a clinical procedure, that lasted for ≥12 h or a >50% reduction in volume over the same time-frame.

SECONDARY OUTCOMES:
Days from birth to full enteral feeding. | Approximately 10 days.
  Full enteral feeding (defined as 150 ml/kg/d).
Number of participants with NEC II-III. | From study day 1 through hospitalization, approximately 60 days.
  NEC II-III defined using Bell's staging criteria with Bell Stage >II classification consisting of clinical symptoms and evidence of septic shock, pneumatosis, bowel perforation, or histologic evidence of bowel ischemia consistent with NEC on bowel resection.
Number of participants with late onset-sepsis. | From study day 1 through hospitalization, approximately 60 days.
  Late-onset sepsis was defined as clinical symptoms and a positive culture in blood, cerebrospinal fluid, or suprapubic or catheter urine ≥5 days post-partum.
Total deaths prior to discharge. | From study day 1 through hospitalization, approximately 60 days.
  Total deaths prior to hospital discharge or discharge from home-care in Sweden.
Number of participants with bronchopulmonary dysplasia. | Assessed at 36 weeks 0 days post-conceptional age.
  Bronchopulmonary dysplasia defined as a need for oxygen support at 36 weeks 0 days.
Number of participants with severe retinopathy of prematurity (ROP). | From study day 1 through hospitalization, approximately 60 days.
  Severe retinopathy of prematurity (ROP) that was treated (e.g. laser or intraocular antivascular injection).

OTHER OUTCOMES:
Cause of death prior to discharge. | From study day 1 through hospitalization, approximately 60 days.
  Cause of death prior to hospital discharge or discharge from home-care in Sweden (exploratory outcome).
Number of participants with surgical NEC. | From study day 1 through hospitalization, approximately 60 days.
  NEC requiring surgical intervention (exploratory outcome).
Mortality and morbidity index. | From study day 1 through hospitalization, approximately 60 days.
  A composite of death, NEC Bell´s II-III, culture-proven sepsis, treated ROP and BPD. (deemed exploratory given a similar composite used as the primary outcome)
Number of withdrawals. | From study day 1 through hospitalization, approximately 60 days.
  Number of infants withdrawn from the intervention for any reason (exploratory outcome).
Days on parenteral nutrition. | Through feeding intervention, approximately 50 days.
  Number of days on parenteral nutrition from birth/from Study Day 1. Defined as receiving amino acids and/or fat intravenously, not just a source of carbohydrate (exploratory outcome).
Percentage of enteral feeds fed as mother's versus PDHM. | Through feeding intervention, approximately 50 days.
  Exploratory outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah L O'Connor, PhD, RN, Principal Investigator — The Hospital for Sick Children; Magnus Domellöf, MD, PhD, Principal Investigator — Umeå University, Umeå (UMU)
Locations (2):
- The Hospital for Sick Children, Toronto, Ontario, Canada
- Umeå University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Data transfer will take place via Secure File Transfer Protocol (SFTP). A sub-agreement which covers data sharing and confidentiality is in place.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: February 2025 to February 2027
Access Criteria: The Hospital for Sick Children (Lead Dr. Deborah L. O'Connor PhD, RD): Data analysis.
  Umeå University - (Lead Dr. Magnus Domellöf MD, PhD): Data analysis.

REFERENCES:
- [Background] Jensen GB, Ahlsson F, Domellof M, Elfvin A, Naver L, Abrahamsson T. Nordic study on human milk fortification in extremely preterm infants: a randomised controlled trial-the N-forte trial. BMJ Open. 2021 Nov 23;11(11):e053400. doi: 10.1136/bmjopen-2021-053400. PMID 34815288
- [Background] Corrigendum for O'Connor et al. Nutrient enrichment of human milk with human and bovine milk-based fortifiers for infants born weighing < 1250 g: a randomized clinical trial. Am J Clin Nutr 2018;108:108-16. Am J Clin Nutr. 2020 May 1;111(5):1112. doi: 10.1093/ajcn/nqaa042. No abstract available. PMID 32367115